CLINICAL TRIAL: NCT06127498
Title: A Randomized, Double-blind, Placebo-parallel Controlled Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of A8G6 COVID-19 Neutralizing Antibody Combination Nasal Spray in Healthy Subjects
Brief Title: The Safety and Tolerability of A8G6 COVID-19 Neutralization Antibody Combined With Nasal Spray
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-69
Record Dates: First submitted 2022-12-27; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2022-12

CONDITIONS: SARS-CoV-2; Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A8G6 SARS-CoV-2 Neutralization Antibody combination nasal spray (Experimental): Specifications: 5 mg/mL, 6 mL/ bottle; Provided by Chongqing Mingdao Haoyue Biotechnology Co., LTD
  Interventions: Biological: A8G6 SARS-CoV-2 Neutralization Antibody combination nasal spray
- A8G6 SARS-CoV-2 Neutralization Antibody nasal excipient (Placebo Comparator): Specification: 0 mg/mL, 6 mL/ bottle; Provided by Chongqing Mingdao Haoyue Biotechnology Co., LTD
  Interventions: Other: A8G6 SARS-CoV-2 Neutralization Antibody nasal excipient

INTERVENTIONS:
Biological: A8G6 SARS-CoV-2 Neutralization Antibody combination nasal spray — Subjects in each cohort were randomly assigned 5:1 to two parallel administration groups, one of which served as a control. Each cohort was given either the experimental drug or placebo by nasal spray at different doses and intervals, and blood was collected on an empty stomach before the first dose. Right nostril and nasal swabs were collected for immunotoxicity, immunogenicity (immunogenicity collection and detection in cohorts 3 and 4 only), and drug concentration detection. Subjects in the first three cohort were required to return to the study Center 3±1 days after the last dose for blood samples, bilateral nostril and nasal swabs for drug concentration, immunotoxicity, physical examination, vital signs, and safety laboratory indicators (blood routine, blood biochemical, and urine routine). Subjects in cohort 4 returned to the study center 7±2 days after the last dose.
  Arms: A8G6 SARS-CoV-2 Neutralization Antibody combination nasal spray
Other: A8G6 SARS-CoV-2 Neutralization Antibody nasal excipient — Subjects in each cohort were randomly assigned 5:1 to two parallel administration groups, one of which served as a control. Each cohort was given either the experimental drug or placebo by nasal spray at different doses and intervals, and blood was collected on an empty stomach before the first dose. Right nostril and nasal swabs were collected for immunotoxicity, immunogenicity (immunogenicity collection and detection in cohorts 3 and 4 only), and drug concentration detection. Subjects in the first three cohort were required to return to the study Center 3±1 days after the last dose for blood samples, bilateral nostril and nasal swabs for drug concentration, immunotoxicity, physical examination, vital signs, and safety laboratory indicators (blood routine, blood biochemical, and urine routine). Subjects in cohort 4 returned to the study center 7±2 days after the last dose.
  Arms: A8G6 SARS-CoV-2 Neutralization Antibody nasal excipient

SUMMARY:
This is a randomized, double-blind, placebo-parallel intervention clinical study that will include approximately 108 healthy subjects based on inclusion and exclusion criteria. Patients meeting inclusion and exclusion criteria were randomly assigned to one of four different cohorts. Subjects in each cohort were randomly assigned 5:1 to two parallel administration groups, one of which served as a control. Each cohort was given either the experimental drug or placebo by nasal spray at different doses and intervals, and blood was collected on an empty stomach before the first dose. Right nostril and nasal swabs were collected for immunotoxicity, immunogenicity (immunogenicity collection and detection in cohorts 3 and 4 only), and drug concentration detection. Subjects in the first three cohort were required to return to the study Center 3±1 days after the last dose for blood samples, bilateral nostril and nasal swabs for drug concentration, immunotoxicity, physical examination, vital signs, and safety laboratory indicators (blood routine, blood biochemical, and urine routine). Subjects in cohort 4 returned to the study center 7±2 days after the last dose. To evaluate the safety and tolerability of A8G6 COVID-19 neutralization and antibody combined nasal spray in healthy subjects by comparing the test results of subjects in different cohorts, and to study its concentration in serum and nasal swabs in healthy subjects.

DETAILED DESCRIPTION:
As of May 11, 2022, more than 519 million COVID-19 cases and 6.28 million deaths have been reported worldwide, according to Worldometer Real-time statistics. On November 27, 2021, a large number of highly transmissible mutated new variants of COVID-19 were found in South Africa, which was named Omicron (including subtypes BA.1 and BA.2) by WHO. Although the introduction of vaccines has played a great role in the prevention and control of COVID-19, the neutralizing antibodies stimulated by different vaccines differ greatly, and the antibody maintains a high titer in the human body for a short time (3-6 months at most), so the global demand for safe and effective prevention of COVID-19 remains unmet.

The novel coronavirus neutralizing antibody can directly bind to the envelope of the novel coronavirus to rapidly block the virus infection, which has been fully verified as a safe and effective treatment. But so far, there are no approved antibodies at home or abroad to prevent infection with the novel coronavirus, In addition, there is a lack of broad-spectrum monoclonal neutralizing antibodies with high efficiency against mutant strains (currently, all the approved neutralizing antibodies in the world are used in combination with two antibodies), which can be used as reference for the administration of neutralizing antibodies for the prevention of a wide range of people (intravenous infusion as the prophylactic administration will lead to low compliance of the administration population).

MY-586 and MY-558, two active components of the novel coronavirus neutralizing antibody A8G6, were screened from peripheral blood lymphocytes of patients recovering from COVID-19, from which 209 strains of novel coronavirus specific antibodies were isolated. The screened MY-586 is a super antibody with strong and effective neutralization against the novel coronavirus and the circulating British strain, Indian strain, South African strain and Indian Delta strain. Its high affinity, high level and activity against the novel coronavirus, broad-spectrum variant strain activity and antibody structure analysis supporting superior activity. It has been published in the authoritative international journal Nature Communications. MY-558 is a super antibody with high affinity, high activity and high affinity to both the novel coronavirus and Omicron (BA.1 and BA.2) strains, and the binding regions of MY-586 and MY-558 and RBD do not overlap, so there is no competitive relationship between the two. On the contrary, the two have certain synergistic effects on each novel coronavirus strain. Among the COVID-19 neutralizing antibodies published worldwide, A8G6 antibody has one of the best affinity and neutralizing activity against COVID-19.

At present, the evaluation of the preclinical efficacy and safety of A8G6 combined antibody and the production of CMC to support the clinic are nearing completion. All the data showed that the A8G6 combined antibody had excellent efficacy, safety and druggability. In particular, A8G6 combined antibody is administered by nasal spray. Although there are no approved nasal spray neutralizing antibody drugs on the market at home and abroad, the investigators have successfully solved the drugging of A8G6 combined antibody by nasal spray and the development of nasal spray device. Nasal spray type A8G6 combined antibody is easy to carry, easy to administer, and has strong accessibility and compliance for the population. It can be used as a new and widely used safe and effective preventive measure besides vaccine. Therefore, the rapid and successful clinical research and development of A8G6 combined antibody will provide a more effective guarantee for social security and effective prevention of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand the purpose, nature, method and possible adverse reactions of the experiment, voluntarily participate in the experiment, and sign informed consent before the experiment begins;
2. Healthy subjects aged 18-65 years (including the critical value) with an appropriate sex ratio between men and women;
3. The subjects had no birth plan for 3 months from the date of signing the informed consent to the end of the study, and agreed to voluntarily take effective and appropriate contraceptive measures with their partners during this period;
4. The subject agrees that from the beginning of the study (-1 day) to the end of the study, except for this study, only samples of NCOV nucleic acid from throat swabs will be taken, and nasal swabs will not be taken;
5. The subjects had not received any type of NCOV vaccine within 3 months prior to enrollment, and had no NCOV vaccination plan during the study period;
6. Subjects can communicate well with researchers and understand and comply with the requirements of this study.

Exclusion Criteria:

1. Allergic to any ingredient in this product and auxiliary materials; Or allergic (such as allergic to two or more drugs, food);
2. Patients with symptoms of acute upper respiratory tract infection within 1 week before administration;
3. Patients with acute episodes of chronic rhinitis or anatomical abnormalities affecting drug absorption in the nose;
4. Patients with a history of asthma;
5. Asplenia or functional asplenia caused by any condition;
6. Diseases or factors with clinical abnormalities that need to be excluded, including but not limited to diseases of the nervous system, cardiovascular system, kidney, liver, gastrointestinal system, respiratory system, metabolism, bone system and other systems;
7. Vital signs, physical examination, laboratory examination (such as white blood cell count less than 3.0*109/L, platelet count less than 75*109/L, TB > 1.5*ULN, ALT > 1*ULN, AST > 1*ULN) and electrocardiogram examination of any items abnormal and judged by the investigator to be clinically significant;
8. Use of any prescription or over-the-counter drugs within 14 days before administration;
9. Patients who had received immunosuppressive therapy, cytotoxic therapy or inhaled corticosteroid therapy within 6 months before administration;
10. A history of drug abuse or use of any drug in the 6 months prior to drug administration;
11. Pregnant and lactating women;
12. The subject has not taken effective and appropriate contraceptive measures within 30 days before the drug administration;
13. The subjects had sperm and egg donation plans within 3 months after the first drug administration to the end of the study;
14. Blood donation or massive blood loss (≥200mL), receiving blood transfusion or using blood products within 3 months prior to drug administration; Or plan to donate blood or blood components during the trial;
15. Have participated in other drug clinical trials or device clinical trials, and have taken test drugs or used test devices within 3 months before drug administration;
16. Subjects may not be able to comply with the protocol to complete the study for other reasons or the investigator may decide that it is not suitable for participants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
vital signs | 14 days before the trial,1 days before the trial, after each dose
  Including pulse, blood pressure, temperature
laboratory tests | 14 days before the trial,1 days before the trial, after each dose
  Including blood routine, blood biochemistry, routine urine pregnancy test (female) limited
12-lead electrocardiogram | 14 days before the trial,1 days before the trial, after each dose
  Including ECG QT Interval、PR Interval
adverse events | Up to 1 year
  Adverse reactions were recorded by questionnaire. Observe any adverse events

SECONDARY OUTCOMES:
Drug concentration index | 15 minutes after each dose
  Serum and nasal swab drug concentration
Immunotoxicity detection indicators | 15 minutes after each dose
  Serum autoantibody titer
Immunogenicity detection indicators | 15 minutes after each dose
  ADA detection of serum MY-586 and MY-558
Cytokines | 15 minutes after each dose
  Serum Cytokines titer
lymphocyte subsets | 15 minutes after each dose
  Serum lymphocyte subsets

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Zhang, M.D., Study Chair — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No